CLINICAL TRIAL: NCT03829397
Title: To Investigate the Correlation of Stroke Patients and Demoralized
Status: Completed | Type: Observational
Sponsor: Taoyuan General Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: TYGH107037
Record Dates: First submitted 2019-01-30; First posted 2019-02-04 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2019-05

CONDITIONS: Post-stroke Depression
Keywords: Demoralization Scale-Mandarin Version; Demoralization syndrome
MeSH Terms: interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Questionnaire — Questionnaire

SUMMARY:
This study aim to clarify the participants's mental state with Demoralization Scale- Mandarin Version(DS-MV). Based on clinical observations and literature review, investigators assume participants's DS-MV score high correlation with PHQ-9 score.

DETAILED DESCRIPTION:
The Chinese version of Demoralization Scale-Mandarin Version (DS-MV) was used to assess the mental state of patients with stroke after debridement. The statistical analysis test of correlation is carried out, and the reliability and validity test and the norm establishment of the Chinese version are further tested. Convenient sampling will be performed at a single medical facility. The planned implementation period is 2019/01/01 ~ 2019/12/31, and the location of the case is the rehabilitation ward and outpatient clinic of Taoyuan Hospital. The diagnosis must be: intensive stroke or hemorrhagic brain within three years. In the case of a 20- to 100-year-old clinical patient with stroke, the subject should explain the content of the case, and the subject will complete the test consent form after informed consent, and then begin the evaluation process of the self-assessment questionnaire. The assessment procedure is preceded by a clinical psychologist conducting with MMSE test to determine the cognitive function. When the patient's consciousness is blurred, the simple intelligent state test (MMSE) score less than 24 points, aphasia can not be effectively communicated, the diagnosis of mental illness or mental disorder has been recorded on the medical record, or the patient or family member is unwilling to sign the informed consent form. If the above situation is met, subjects will be excluded. The self-assessment questionnaire will obtain the scores of the subjects in the Chinese version of the Demoralization Scale-Mandarin Version (DS-MV) and the Patient Health Questionnaire (PHQ-9). Statistical analysis, as well as the Chinese version of the loss of the scale of the reliability and validity of the test and the establishment of clinical norm scores.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient and outpatient of rehabilitation department in Taoyuan General Hospital, patients diagnosis : who have an infarct stroke or hemorrhagic stroke within three years.

Exclusion Criteria:

* Conscious state confusion, the MMSE score less than 24.
* Unable to understand information, speech disorders, dementia, aphasia.
* The diagnosis of mental illness or mental disorder has been recorded on the medical history.
* The patient or family unwilling to sign an informed consent.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: infarct stroke or hemorrhagic stroke within three years
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
demoralization Scale-Mandarin Version (DS-MV) total score | through study completion, an average of 1 year
  When participants was included, investigators get on one-time assessment use the demoralization Scale-Mandarin Version (DS-MV). The demoralization Scale-Mandarin Version (DS-MV) minimum score are 0, and maximum score are 96, cut-off point are 30. No subscale.

SECONDARY OUTCOMES:
demoralization Scale-Mandarin Version (DS-MV) total score split-half reliability | through study completion, an average of 1 year
  Divide the demoralization Scale-Mandarin Version (DS-MV) into half, and then test the items of the previous half (item 1-12) and the second half (item 13-24) of the questionnaire. Then the two half questionnaire scores were test of correlation coefficient.Then If the degree of correlation is high, the reliability is very high.
Patient Health Questionnaire (PHQ-9) total score | through study completion, an average of 1 year
  When participants was included, investigators get on one-time assessment use the Patient Health Questionnaire (PHQ-9) .Patient Health Questionnaire (PHQ-9) minimum score are 0, and maximum score are 27. No subscale.
demoralization Scale-Mandarin Version (DS-MV) total score criterion-related validity | through study completion, an average of 1 year
  Correlation test between demoralization Scale-Mandarin Version (DS-MV) total score and Patient Health Questionnaire(PHQ-9) total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Tao-Yuan General Hospital, Taoyuan, Zhongshan Rd., Taoyuan Dist, Taiwan

REFERENCES:
- [Background] Nanni MG, Caruso R, Travado L, Ventura C, Palma A, Berardi AM, Meggiolaro E, Ruffilli F, Martins C, Kissane D, Grassi L. Relationship of demoralization with anxiety, depression, and quality of life: A Southern European study of Italian and Portuguese cancer patients. Psychooncology. 2018 Nov;27(11):2616-2622. doi: 10.1002/pon.4824. Epub 2018 Aug 6. PMID 29943491
- [Background] Tang PL, Wang HH, Chou FH. A Systematic Review and Meta-Analysis of Demoralization and Depression in Patients With Cancer. Psychosomatics. 2015 Nov-Dec;56(6):634-43. doi: 10.1016/j.psym.2015.06.005. Epub 2015 Jun 19. PMID 26411374
- [Background] Juliao M, Nunes B, Barbosa A. Prevalence and factors associated with demoralization syndrome in patients with advanced disease: Results from a cross-sectional Portuguese study. Palliat Support Care. 2016 Oct;14(5):468-73. doi: 10.1017/S1478951515001364. Epub 2016 Jan 6. PMID 26732616
- [Background] Wu YC, Tung HH, Wei J. Quality of life, demoralization syndrome and health-related lifestyle in cardiac transplant recipients - a longitudinal study in Taiwan. Eur J Cardiovasc Nurs. 2019 Feb;18(2):149-162. doi: 10.1177/1474515118800397. Epub 2018 Sep 18. PMID 30226074
- [Result] Clarke DM, Kissane DW. Demoralization: its phenomenology and importance. Aust N Z J Psychiatry. 2002 Dec;36(6):733-42. doi: 10.1046/j.1440-1614.2002.01086.x. PMID 12406115
- [Result] Mangelli L, Semprini F, Sirri L, Fava GA, Sonino N. Use of the Diagnostic Criteria for Psychosomatic Research (DCPR) in a community sample. Psychosomatics. 2006 Mar-Apr;47(2):143-6. doi: 10.1176/appi.psy.47.2.143. PMID 16508026
- [Result] Robinson S, Kissane DW, Brooker J, Burney S. A systematic review of the demoralization syndrome in individuals with progressive disease and cancer: a decade of research. J Pain Symptom Manage. 2015 Mar;49(3):595-610. doi: 10.1016/j.jpainsymman.2014.07.008. Epub 2014 Aug 15. PMID 25131888